CLINICAL TRIAL: NCT01059526
Title: A Phase 4, Long-Term Observational Safety Study to Evaluate Immunogenicity and Hypersensitivity With Exposure to KALBITOR (Ecallantide) for the Treatment of Acute Attacks of HAE
Brief Title: Observational Safety Study for KALBITOR (Ecallantide) in the Treatment of Acute Attacks of Hereditary Angioedema
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: DX-88/24
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — ecallantide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients naive to KALBITOR: HAE patients that have not been treated with KALBITOR (ecallantide) prior to enrollment in the study
  Interventions: Drug: ecallantide
- Patients non- naive to KALBITOR: HAE patients that have been treated with KALBITOR prior to enrollment in the study
  Interventions: Drug: ecallantide

INTERVENTIONS:
Drug: ecallantide — 30 mg SC
  Other Names: Kalbitor

SUMMARY:
The objective of this study is to evaluate the formation of antibodies, the occurence of allergic reactions, and the risk of hypercoagulability and hypocoagulability in patients treated with KALBITOR (ecallantide).

DETAILED DESCRIPTION:
The objective of this study is to evaluate immunogenicity and hypersensitivity upon exposure to KALBITOR, in particular:

1. Determine the rate of anaphylaxis and Type I hypersensitivity reactions upon exposure to KALBITOR.
2. Determine the rate of seroconversion to anti-ecallantide antibodies upon exposure to KALBITOR.
3. Determine the rate of adverse events related to disordered coagulation (hypercoagulability and hypocoagulability) upon exposure to KALBITOR.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated per the approved product label for KALBITOR
* Patient or guardian is able to understand and sign the informed consent form
* Patient is willing and able to undergo a skin test procedure at screening (baseline)

Exclusion Criteria:

* Patient contraindicated per the approved product label for KALBITOR
* Patient confirmed pregnancy or active breastfeeding
* Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful completion of the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hereditary angioedema, either naive or non-naive to KALBITOR (ecallantide) prior to enrollment in the study
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2014-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (40):
- United States (40):
  - Little Rock Allergry and Asthma Clinical Research Center, Little Rock, Arkansas
  - Sunrise Clinical Research, Bell Gardens, California
  - Allergy & Asthma Institute of the Valley, Granada Hills, California
  - Unidversity of California, Los Angeles David Geffen School of Medicine, Los Angeles, California
  - 705 West LaVeta, Orange, California
  - Allergy & Asthma Clinical Research Inc., Walnut Creek, California
  - Center for Allergy, Asthma & Immunology, Waterbury, Connecticut
  - University of South Florida Asthma, Tampa, Florida
  - Brookstone Clinical Research Center, Columbus, Georgia
  - University Consultants in Allergry and Immunology, Chicago, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Muncie Allergy Ctr, Muncie, Indiana
  - Kansas City Allergy and Asthma Associates, Overland Park, Kansas
  - Ochsner Health System - Allergy, Asthma and Immunology Department, Jefferson, Louisiana
  - Clinical Research Specialists, Metairie, Louisiana
  - Institute for Asthma and Allergy, P.C., Chevy Chase, Maryland
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - University of Michigan Health System Allergy Specialty Clinic, Ann Arbor, Michigan
  - Asthma and Allergy Institute of Michigan, Clinton Township, Michigan
  - Saint Louis University School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nevada School of Medicine - Department of Pediatrics, Reno, Nevada
  - Allergy Treatment Center of New Jersey, Iselin, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Medical Research Associates of CNY, North Syracuse, New York
  - The Bronx, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Specialty Medical Clinic And Research Center, Sanford, North Carolina
  - Department of Internal Medicine, University of Cincinnati -MSB, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Reynolds Clinic, Toledo, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Allergy Clinic of the Tulsa, Inc., Tulsa, Oklahoma
  - Penn State University - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - University of Utah, Department of Dermatology, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Virginia Beach, Virginia
  - Puget Sound Allergy, Asthma and Immunology, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients indicated in the US FDA-approved product label for KALBITOR (ecallantide) who experienced an acute attack of HAE were eligible for inclusion in this trial.
Pre-assignment Details: Subjects were to complete screening/enrollment procedures on a separate day prior to receiving KALBITOR treatment for an acute attack of HAE. The primary and secondary endpoints were analyzed for the Safety population only (all patients who received at least 1 treatment dose of KALBITOR).
Groups:
- Patients Naive to KALBITOR: HAE patients that have not been treated with KALBITOR (ecallantide) prior to enrollment in the study ecallantide: 30 mg SC
- Patients Non- Naive to KALBITOR: HAE patients that have been treated with KALBITOR prior to enrollment in the study ecallantide: 30 mg SC
Period: Overall Study
Arm/Group | Patients Naive to KALBITOR | Patients Non- Naive to KALBITOR
Started | 41 (ITT population; defined as signing informed consent and meeting all inclusion/ exclusion criteria) | 40 (ITT population; defined as signing informed consent and meeting all inclusion/ exclusion criteria)
Treated | 21 (Safety population; defined as all patients who received at least 1 treatment dose of KALBITOR) | 23 (Safety population; defined as all patients who received at least 1 treatment dose of KALBITOR)
Completed | 11 | 18
Not Completed | 30 | 22
Not completed — Patient enrolled but not treated | 20 | 17
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Patient found to be dermatographic | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population; defined as all patients who received at least 1 treatment dose of KALBITOR
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Naive to KALBITOR | Patients Non- Naive to KALBITOR | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (16.09) | 38.3 (14.86) | 43.0 (16.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 6 | 8 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20 | 22 | 42
  Black | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Anaphylaxis or Other Adverse Events Suggestive of Hypersensitivity
Description: Based on medical review of multiple preferred terms for treatment emergent adverse events (TEAEs) suggestive of Type 1 hypersensitivity; terms included adverse drug reaction, anaphylaxis, anaphylactic reaction, anaphylactoid reaction, hypersensitivity, erythema, flushing, hot flush, pharyngeal edema, laryngeal edema, pruritus, pruritus generalized, rash, rash erythematous, rhinitis allergic, rhinorrhea, throat irritation, urticaria, urticaria localized, dyspnea, and wheezing. Records of patients with any of these TEAE referred terms were reviewed further to assess potential hypersensitivity reactions, considering factors such as timing of TEAEs in relationship to dose (ie, occurred within 24 hours after start of KALBITOR treatment), accompanying symptoms, Investigator causality assessment (ie, reported as possibly, probably, or definitely related to study drug), and any other available clinical information. Anaphylaxis subset determined based on criteria established by the NIAID.
Time Frame: 12 months after first treatment
Population: Safety population; defined as all patients who received at least 1 treatment dose of KALBITOR
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Safety Population: Safety population; defined as all patients who received at least 1 treatment dose of KALBITOR
Arm/Group | Safety Population
Number analyzed (Participants) | 44
participants
  Type 1 hypersensitivity | 4 [0.6 to 17.6]
  Anaphylaxis per NIAID criteria | 2 [0.0 to 10.7]

2. Primary Outcome: Occurrence of Seroconversion to Anti-ecallantide Antibodies Upon Exposure to KALBITOR.
Description: Seroconversion is the development of detectable specific antibodies in the blood serum. Serum was tested for development of antibodies (irrespective of immunoglobulin class) against ecallantide at screening and at all safety evaluations. Positive results were to undergo a confirmatory test. Confirmed positive samples were further titered. Patients who developed an antibody response were evaluated for the development of neutralizing antibodies. Patients also had their serum analyzed for IgE-specific antibodies to ecallantide at screening and during safety evaluations. Positive results underwent a confirmatory test. Confirmed positive samples were further titered.
Time Frame: 12 months after first treatment
Population: Based on total number of patients who were not positive for the antibody class at study entry and had at least one post-baseline antibody evaluation. N=40 evaluable patients for all immunoglobulin antibody classes; N=41 evaluable patients for IgE to ecallantide antibodies; N=41 evaluable patients for neutralizing antibodies to ecallantide.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 41
participants
  Seroconversion based on all Ig antibody classes | 6 [3.9 to 26.1]
  Seroconversion based on IgE to ecallantide | 0 [NA to NA] — NA = 95% CI is not evaluable for 0 events
  Seroconversion based on neutralizing antibodies | 5 [2.2 to 22.2]

3. Primary Outcome: Occurrence of Adverse Events Related to Disordered Coagulation (Hypercoagulability and Hypocoagulability) Upon Exposure to KALBITOR
Description: Events of ecchymosis, hemorrhage, petechiae, spontaneous hemorrhage, hematoma, gastrointestinal bleeding, hemorrhagic stroke and any other term indicative of a bleeding event or increased tendency for bleeding were reviewed to determine the occurrence of hypocoagulability. Events of clotting, thrombosis, pulmonary embolism, vaso-occlusive stroke, myocardial infarction, and any other term indicative of a clotting event or increased risk of clotting were reviewed to determine the occurrence of hypercoagulability.
Time Frame: 12 months after first treatment
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Safety Population
Number analyzed (Participants) | 44
participants | 0 [NA to NA] — NA = 95% CI is not evaluable for 0 events

4. Secondary Outcome: Overall Patient Response Assessment
Description: The Overall Response Assessment was to be completed every 30 minutes after treatment until patient discharge. Patients evaluated their response to treatment as "a lot better or resolved," "a little better," "the same," "a little worse," or "a lot worse." The data presented is based on the best response achieved following a single dose of KALBITOR (Dose A) for the first HAE treatment episode. Responses of "a lot better or resolved" and "a little better" were combined to form a category of "Better." Similarly, "a little worse" and "a lot worse" were combined to form a category of "Worse." Patients treated in a clinic (study site) could have been discharged after an hour and hence may have only had 2 post-treatment evaluations (30 and 60 minutes); response assessments may not have been consistently provided when patients were treated at an alternate site outside of the study site.
Time Frame: within 4 hours post dose
Population: Safety population; defined as all patients who received at least 1 treatment dose of KALBITOR. Analysis only includes episodes of patients who were treated at the study site.
Measure: Number; unit: participants
Arm/Group | Patients Naive to KALBITOR | Patients Non- Naive to KALBITOR
Number analyzed (Participants) | 11 | 17
participants
  Better | 10 | 15
  Same | 1 | 2
  Worse | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months after first treatment
Description: Adverse events were to be recorded for the duration of the study. Results are presented for episode-based treatment-emergent adverse events--ie, those that occurred or worsened in severity within 24 hours after the start of treatment with KALBITOR, or were reported as related to treatment with KALBITOR regardless of time of onset post treatment.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 6/44
Other Adverse Events (participants affected / at risk) | 14/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=44)
Dehydration (Metabolism and nutrition disorders) | 2
Hereditary angioedema (Congenital, familial and genetic disorders) | 2
Drug ineffective for unapproved indication (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=44)
Skin test positive (Investigations) | 5
Hereditary angioedema (Congenital, familial and genetic disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
44 patients (out of 200 planned) received treatment in this study. Additionally, the collection of evaluable efficacy data for the secondary endpoint was limited by a lack of response data collected for HAE attacks treated at alternate sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dyax agreements vary, but Dyax will not prohibit any investigator from publishing. Dyax reviews publications prior to public release and can request deferral by up to 60 days beyond the proposed publication date if necessary to preserve its intellectual property. Dyax can request changes to publications to remove non-study-related confidential information. Dyax can also request deferral of single-center publications until after disclosure of the clinical trial's primary publication.